CLINICAL TRIAL: NCT04778306
Title: Comparision of Oncological Results of Transoral Laser Surgery and Radiotheraphy for Early Stage Laryngeal Squamous Cell Cancer: Single Center Median Long-term Results.
Brief Title: Transoral Laser Surgery and Radiotheraphy for Early Stage Laryngeal Squamous Cell Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Sumeyra DOLUOGLU, Principal Investigator, Saglik Bilimleri Universitesi
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SBUADYBTRH
Record Dates: First submitted 2021-02-21; First posted 2021-03-03 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-02

CONDITIONS: Larynx Cancer
Keywords: Early stage laryngeal cancer; Oncological results; Squamous cell laryngeal cancer
MeSH Terms: conditions — Laryngeal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trans Oral Laser Surgery (Group 1) (Active Comparator): In TOLS, the tumor tissue was removed en bloc and in one piece. The removed specimen was marked on a card with the help of pins. Permanent surgical margins were taken from the anterior, posterior, superior, inferior and deep areas of the tumor area.
  Interventions: Procedure: Transoral Laser Surgery
- Radiotherapy (Group 2). (Active Comparator): . In RT; the head was routinely stabilized with the help of a thermoplastic mask and subsequently covered the primary area with a size varying from 4x4 cm to 6x6 cm. Total 63-70 Gy radiotherapy was applied 2.0-2.3 Gy/ day,5 days a week, for 6-7 weeks.
  Interventions: Procedure: Transoral Laser Surgery

INTERVENTIONS:
Procedure: Transoral Laser Surgery — Remove of the laryngeal tumour via diode laser

SUMMARY:
Background: The investigators aimed to compare the oncological results of patients with early stage laryngeal squamous cell carcinoma (LSCC) treated with Transoral Laryngeal Surgery (TOLS) and Radiotheraphy (RT).

Methods: The patients were divided into two groups as TOLS (Group 1) and RT (Group 2) according to the treatment method. Both groups were compared with each other in terms of local recurrence, regional recurrence, distant metastasis, 3 and 5-year overall survival, disease-free survival, disease-specific survival and laryngectomy-free survival rates. Survival analyses was made by Kaplan Meier product limit estimation. A p-value of less than 0.05 was considered as statistically significant.

DETAILED DESCRIPTION:
Laryngeal cancers are one of the most common head and neck cancers (HNC). According to the 2018 cancer statistics, the estimated number of new laryngeal cancer cases annually is 177.000, and approximately half of these cases died due to the laryngeal cancer. While the most common HNC in the world is oral cavity cancer, in Turkey the most common HNC is laryngeal cancer. In Turkey, laryngeal cancers are showed 6.6/ 100.000 in men, 0.5/ 100.000 in women, and it ranked eighth in cancer deaths in men. Every year in Turkey, more than 3500 cases of new laryngeal cancer are expected, and its incidence has increased significantly in the last ten years.

In the main treatment of early stage laryngeal cancers, surgery (transoral laryngeal surgery (TOLS) - open partial laryngeal surgery (OPLS)) and radiotherapy (RT) are used. Although the oncological results of all of three treatment strategies are similar, TOLS performed with laser is preferred mostly because of short hospital stay, low cost, good functional result, low morbidity and mortality.

There are quite different studies in the literature on whether surgical and non-surgical treatment methods used in the treatment of early stage laryngeal cancers are superior to each other in terms of oncological results. In a randomized controlled study with a large patient series comparing surgery and radiotherapy, 5-year overall survival (OS) in T1 tumors (91.7% in the RT group, 100% in the surgery group) and in T2 tumors (88.8% in the RT group, 97.4% in the surgery group) was similar. 5-year disease-free survival (DFS) in T2 tumors (60.1% in RT group, 78.7% in surgery group) was higher in favor of surgery. Studies comparing TOLS and radiotheraphy in the treatment of early stage laryngeal cancer within the last 20 years have reported comparable oncologic outcomes; two recent meta-analyses have reported better overall survival after TOLS than radiotheraphy, despite being able to show any difference in local control. In this study, we aimed to compare the effects of TOLS and RT on local control, regional control, overall survival (OS), disease-free survival (DFS), disease-specific survival (DSS) and larynjectomy-free survival (LFS) in early stage laryngeal cancers in our own series of patients with high patient volume and long follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Early stage laryngeal cancer (Tis-1-2N0M0)
* >18 years old.

Exclusion Criteria:

* <18 years old
* History of another malignant disease
* Incomplete data
* Non-squamous cell carcinoma
* No follow-up.

Ages: 33 Years to 83 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 261 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Overall survival | at least 1 year
  Overall survival

IPD SHARING:
Plan to Share IPD: No